CLINICAL TRIAL: NCT06025721
Title: Development of a Multiple Health Behavior Change Intervention for Cardiovascular Risk Reduction Among People Who Have Experienced Homelessness: The CV-HOMES Study
Brief Title: Behavior Change Intervention for Cardiovascular Risk Reduction Among People Experiencing Homelessness
Acronym: CV-Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katherine Vickery (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Minnesota (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor-Investigator, Katherine Vickery, Katherine Vickery, MD, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2022-373; P50MD017342 (NIH)
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Heart Diseases; Diabetes Mellitus, Type 2; Pre-diabetes; Hypertension; Hyperlipidemias
Keywords: Cardiovascular Health; Homeless persons; Delivery of Health Care, Integrated; Primary care; Social determinants of health
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus, Type 2; Glucose Intolerance; Hypertension; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: This will be an in-person, phone, or video based behavioral intervention. It will involve a wellness coach assisting participants to set goals related to diabetes self-care and co-morbitities or social conditions that get in the way of health and wellness. There will be encouragement to work on medication adherence and to address getting healthy sleep, quitting tobacco, being more active, and eating better.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CV-Homes Intervention (Experimental): Behavioral treatment by a wellness coach.
  Interventions: Behavioral: Cardiovascular Risk Homeless Support

INTERVENTIONS:
Behavioral: Cardiovascular Risk Homeless Support — There will be 10 sessions offered within 12 weeks to participants. Sessions will last 30-60 minutes. During sessions a wellness coach will use behavioral activation and motivational interviewing to get to know participants and set goals to improve cardiovascular health behaviors. The coach will encourage a focus on smoking>medication>sleep>physical activity>healthy eating to the extent that participants are willing. The coach will also help with resources and care coordination. The coach will also provide brief cardiovascular health education as needed in participants' preferred format (handout, video, audio, etc.).
  Other Names: CV-Homes

SUMMARY:
This single-arm trial of the Cardiovascular Risk Reduction Among People Experiencing Homelessness (CV-Homes) intervention alone (n=8) will test the perception and feasibility of anticipated study procedures.

DETAILED DESCRIPTION:
This study is of a set of studies with an overall goal to develop and pilot test a collaborative care intervention using motivational interviewing and behavioral activation alongside education and psychosocial support to improve medication adherence tailored to the experiences of people experiencing homelessness and cardiovascular health risks (CV-H). Our team's central hypothesis is that medication adherence and cardiovascular self-care (and eventual glycemic control, cholesterol control, health care use/cost) will improve with an intervention tailored to the unique context of CV-H.

This protocol addresses a pilot study to test patient perceptions of the feasibility and acceptability of study procedures and refine the CV-Homes treatment manual through test cases (n=8). With a hypothesis that the CV-Homes manual and study procedures will be feasible and acceptable to CV-H as measured by self-report and post-treatment interview.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 yrs. or older
* English-speaking
* Living at Catholic Charities' Endeavors residence (Minneapolis, MN)
* Self-reported diagnosis of moderate or high CVD risk, defined as being told by a medical professional that the participant has hypertension, heart disease, hypercholesterolemail, prediabetes, or type 2 diabetes
* Plan to stay in local area or be reachable by phone for the next 16 weeks
* Willingness to work on one or more CVD risk reduction behavior change

Exclusion Criteria:

* Active intoxication
* Active psychosis
* Presence of a legal guardian
* Pregnant or lactating people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Vickery, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin Healthcare Research Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lloyd-Jones DM, Allen NB, Anderson CAM, Black T, Brewer LC, Foraker RE, Grandner MA, Lavretsky H, Perak AM, Sharma G, Rosamond W; American Heart Association. Life's Essential 8: Updating and Enhancing the American Heart Association's Construct of Cardiovascular Health: A Presidential Advisory From the American Heart Association. Circulation. 2022 Aug 2;146(5):e18-e43. doi: 10.1161/CIR.0000000000001078. Epub 2022 Jun 29. PMID 35766027
- [Background] Gathright EC, Vickery KD, Ayenew W, Whited MC, Adkins-Hempel M, Chrastek M, Carter JK, Rosen RK, Wu WC, Busch AM. The development and pilot testing of a behavioral activation-based treatment for depressed mood and multiple health behavior change in patients with recent acute coronary syndrome. PLoS One. 2022 Feb 3;17(2):e0261490. doi: 10.1371/journal.pone.0261490. eCollection 2022. PMID 35113860

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CV-Homes Intervention
Started | 9
Completed | 6
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1
Not completed — Incarceration | 1

BASELINE CHARACTERISTICS:
Arm/Group | CV-Homes Intervention
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Acceptability Measured by the Client Satisfaction Questionnaire
Description: This will be assessed at the end of the intervention using the 8-item Client Satisfaction Questionnaire, with a score range 8-32, higher score indicating greater satisfaction.
Time Frame: at 16 weeks
Population: One participant did not complete the final assessment and one participant skipped this section.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | CV-Homes Intervention
Number analyzed (Participants) | 5
score on a scale | 31 [30 to 32]

2. Primary Outcome: Treatment Engagement Measured by Sessions Attended
Description: Throughout the study we will measure engagement by tracking attendance of treatment sessions.
Time Frame: At 16 weeks
Measure: Mean (Full Range); unit: sessions attended
Arm/Group | CV-Homes Intervention
Number analyzed (Participants) | 7
sessions attended | 6.8 [4 to 10]

3. Secondary Outcome: Health-related Quality of Life
Description: Health related quality of life as measured by the Euro-Qol 5D-5-L which asks 5 questions on a 5-response likert scale with 1 = no problems and 5= unable to, shared as a mean total of responses to the 5 questions with lower scores being higher quality of life and higher scores being lower quality of life. The highest possible score for the 5 questions on the 5-response likert scale (the sum of each response) is 25 and the lowest score is 5. The Euro-Qol also includes one question on a scale of 1-100 with 1 being the worst health one can imagine and 100 being the best health one can imagine.
Time Frame: Baseline to 16 weeks
Population: Baseline included participants who completed baseline survey and began coaching. 16 weeks included participants who completed final assessment.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | CV-Homes Intervention
Number analyzed (Participants) | 7
units on a scale
  5-response scale Baseline | 11.7 [7 to 16]
  5-resonse scale 16 weeks: number analyzed (Participants) | 5
  5-resonse scale 16 weeks | 10.2 [6 to 19]
  1-100 scale Baseline | 58.6 [35 to 75]
  1-100 scale 16 weeks: number analyzed (Participants) | 5
  1-100 scale 16 weeks | 65 [44 to 78]

4. Secondary Outcome: Cardiovascular Health (AHA Life's Essential 8)
Description: Composite measure of self-reported behaviors (healthy eating, physical activity, tobacco use, sleep) and biometric measures (BMI, Blood pressure, Cholesterol, HbA1c). Score is 0-100 with higher scores meaning better cardiovascular health.
Time Frame: Baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CV-Homes Intervention
Number analyzed (Participants) | 6
score on a scale
  Baseline | 52.92 (10.73)
  Final Assessment | 55.52 (9.74)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entire 16 weeks of each participant's involvement in the study.
Arm/Group | CV-Homes Intervention
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT06025721/Prot_SAP_000.pdf